CLINICAL TRIAL: NCT04985175
Title: Impact of Decision Quality by Using Question Prompt List on the Shared Decision Making in End-stage Renal Disease Patients
Brief Title: Impact of Decision Quality by Using Question Prompt List
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 202104009RINA
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-05

CONDITIONS: Decision Making
Keywords: Question prompt list; Shared decision making; End-stage renal disease; Health literacy
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: Subjects were randomized assigned to QPL group or usual care group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QPL group (Experimental): receive 2-pages ESRD QPL leaflets, circle the questions they want to ask before consultation. encourage asking questions with doctor during consultation. receive the nurse-led coaching of shared decision-making (SDM)
  Interventions: Behavioral: Question prompt list
- Usual care group (No Intervention): without receiving provision of QPL encourage asking questions with doctor during consultation. receive the nurse-led coaching of shared decision-making (SDM)

INTERVENTIONS:
Behavioral: Question prompt list — The specific QPS was a one page leaflet for chronic kidney disease which developed by applied literature and public QPL from the National Health Agency. It contains 3 domains 25 questions related to treatment, dialysis, and Kidney transplant. The QPL group participants were asked to read and mark those questions they concerned or write down additional problems.
  Arms: QPL group

SUMMARY:
To investigate the effects of a question prompt list (QPL) on a shared decision-making consultation among facing decision for dialysis in end-stage renal disease (ESRD) patients. A randomized controlled trial was conducted at the university medical center of North Taiwan. Subjects were randomized assigned to QPL group or usual care group. Decisional quality and decision control preferences were assessed with questionnaires. Measurements were performed at before the counseling (T0), immediately after counseling (T1), and evaluate decision regret at one month after treatment.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effectiveness of decisional quality and decisional control preferences by using a specific question prompt list (QPL) during a shared decision-making consultation among facing decision for dialysis in end-stage renal disease (ESRD) patients. A randomized controlled trial was conducted at the university medical center of North Taiwan. Recruit subjects are those who are about to receive the nurse-led coaching of shared decision-making (SDM) for patients with ESRD and attend the program. By using blocked Randomization design, the investigators assigned participants to QPL group or usual care. Prior to a clinic visit to discuss treatment, two-pages ESRD QPL leaflets are provided to QPL group, while usual care group without receiving provision of QPL. Measurements of outcome included decision quality (decision conflict, decisional self-efficiency) and decision control preference at before the counseling (T0), immediately after counseling (T1), and evaluate decision regret at one month after treatment (T2), at this time the patient has decided and started to accept the selected treatment (hemodialysis, peritoneal dialysis or conservative treatment). All statistical analyses were performed in SAS statistical software, version 9.4 (SAS, Cary, NC). The effects of the intervention were assessed by generalized estimating equation (GEE) analysis with the coefficient of interaction ( group × time) term. Statistical tests were two-sided with a significance level of 0.05. Hierarchical Linear Model was used to detect the impact of nested within physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage 5 chronic kidney disease who facing decision for dialysis;
* normal cognitive functions;
* be able to read, communicate in Mandarin or Taiwanese;
* ability to express willingness;

Exclusion Criteria:

* vision or hearing function impairment;
* Severe illness;
* Urgent to dialysis for extend life;
* Dialysis modalities Already decided.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2021-08-15 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Decision conflict | before the counseling (T0), immediately after counseling(T1)
  Decision conflict was measured by Decision conflict scale(DCS). The scale consists of 16 items into 5 subscales: Uncertainty(3 items), Informed(3 items), values clarity(3 items), support(3 items), and effective decision(4 items) that are rated on a 5-point likert-scale from "strongly agree" (0) to "strongly disagree" (4). The sum of scores are calculated from 0 to 100. The higher the score, the higher the level of decision conflict.
Decisional self-efficiency | before the counseling (T0), immediately after counseling(T1)
  Decision self-efficiency was measured by Decisional Self-Efficiency Scale(DSES). The scale represents self-confidence or belief in decision making. The scale consists of 11 items that are rated on a 5-point likert-scale from "not at all confident" (0) to" very confident "(4) . The sum of scores are calculated from 0 to 100. The higher the score, the higher the level of self-confidence.

SECONDARY OUTCOMES:
Decision control preference | one month after treatment (T2)
  Decision regret was measured by Decision regret Scale(DRS) .The scale consists of 5 items that are rated on a 5-point likert-scale from "strongly agree "(1) to" strongly disagree" (5) . The sum of scores are calculated from 0 to 100. The higher the score, the higher the level of regret.
Decision control preference | before the counseling (T0), immediately after counseling(T1)
  Decision control preference was measured by Decision control preference Scale(DCPS) .The scale asks two question:(1)control preference measured at before the counseling; (2) actual decision control level measured after counseling immediately.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Xindian, Taiwan